CLINICAL TRIAL: NCT04989296
Title: Informative Value of Determining the Level of NF-κB Translocation by Flow Cytometry With Visualization in Lymphocyte Populations in Children With Psoriasis
Brief Title: Informative Value of Determining the Level of NF-κB Translocation in Lymphocyte Populations in Children With Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Children's Health, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 05912657
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis Vulgaris
Keywords: NF-κB translocation; Lymphocytes; Flow cytometry with imaging (Amnis); Biological drugs; Сhildren and adolescents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Level of NF-κB translocation in lymphocyte in children with psoriasis and in comparison group (Experimental): The analysis of the relative count of cells with NF-κB translocation in the lymphocyte populations the group of patients with psoriasis and in the comparison group.
  Interventions: Diagnostic Test: Peripheral blood samples were obtained following the standard procedures.
- Level of NF-κB translocation in lymphocyte in children with psoriasis, based on the type of therapy (Experimental): Determination of the level of NF-kB translocation in lymphocyte populations in patient groups depending on the type of therapy: Group 1 - patients receiving basic and external therapy; Group 2 - patients receiving methotrexate; and Group 3 - patients receiving therapy with biological drugs.
  Interventions: Diagnostic Test: Peripheral blood samples were obtained following the standard procedures.
- Severity of psoriasis based on level of NF-κB translocation in psoriasis who received biologics (Experimental): Assessment of the level of NF-kB translocation in lymphocyte populations, assessment of PASI and BSA, assessment of the effectiveness of biological drugs in patients with psoriasis. Identification of patients in the stage of regression of the disease and in the progressive stage.
  Interventions: Diagnostic Test: Peripheral blood samples were obtained following the standard procedures.

INTERVENTIONS:
Diagnostic Test: Peripheral blood samples were obtained following the standard procedures. — Taking 4 ml of peripheral blood from patients on an empty stomach.

SUMMARY:
This study is the first to quantify the level of NF-kB translocation in lymphocyte populations in children and adolescents with psoriasis of varying severity.

DETAILED DESCRIPTION:
This is a diagnostic study aimed at finding immunological predictors of the effectiveness of therapy in children and adolescents with psoriasis.

The study included 90 patients from 1 to 18 years old with psoriasis vulgaris, mild / moderate and severe. The comparison group consisted of 30 healthy children.

The study took into account the PASI (Psoriasis Area Severity Index); the BSA (Body Surface Area); including patient age; duration of the disease; type of therapy; duration of therapy. Depending on the type of therapy, all psoriatic children were divided into 3 groups: Group 1 (n = 24) - patients receiving basic and external therapy; Group 2 (n = 20) - patients receiving systemic therapy with methotrexate; and Group 3 (n = 46) - patients receiving therapy with genetically engineered biological drugs (Adalimumab, Etanercept, Ustekinumab).

The analysis of the NF-κB translocation level in lymphocytes was performed by flow cytometry with imaging (Image Stream Mark II - AMNIS) using the Amnis NF-κB Translocation Kit.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 1 to 18 years old
2. Mild, moderate, and severe psoriasis
3. Healthy children, as a comparison group
4. Patients receiving basic and external therapy, receiving systemic therapy with methotrexate and patients receiving therapy with biological drugs (Adalimumab, Etanercept, Ustekinumab)
5. A signed and dated informed consent received from the patient's parents (guardians), as well as from a patient over 14 years of age, to participate in the study
6. Ability to attend control visits within the specified time frame

Exclusion Criteria:

1. The presence of other concomitant skin diseases in the present or in the past, which could affect the assessment of the effect of the study drugs on the course of psoriasis
2. Use of other genetically engineered biological preparations in therapy
3. Participation in other clinical trials
4. Extensive or complete disability, significantly limiting personal care or determining the inability to carry it out
5. Immunodeficiency disease
6. The presence in the past or present of any serious and / or unstable concomitant disease
7. The course of a viral, bacterial, fungal or parasitic infection

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
The level of NF-kB translocation in lymphocyte populations | Screening on the 1 day of blood sampling
  Changes in NF-kB translocation in lymphocyte populations
Patient age | from 1 to 18 years old
  Age assessment
PASI (Psoriasis Area Severity Index) | 1 day Screening at the time of examination
  Change of the PASI
BSA (Body Surface Area) | 1 day Screening at the time of examination
  Assessment of the affected area of the patient's body

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Children's Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided